CLINICAL TRIAL: NCT02060942
Title: Mean Systemic Filling Pressure and Heart Performance as Predictors of Successful Fluid Responsiveness in Patients With Coronary Artery Bypass Grafting
Brief Title: Mean Systemic Filling Pressure and Heart Performance Predicting Fluid Responsiveness
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, L.P.B. Meijs, MD, PhD-candidate Intensive Care Unit / resident cardiology, Catharina Ziekenhuis Eindhoven
Other Study IDs: M12-1271
Record Dates: First submitted 2013-08-23; First posted 2014-02-12 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Output, High
Keywords: Volume responsiveness mean systemic filling pressure
MeSH Terms: conditions — Cardiac Output, High

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary artery bypass grafting: Post Anaesthetic Care Unit (PACU) patients treated with coronary artery bypass grafting (CABG) are highly eligible for this study. These are patients with an indication for fast track treatment (PACU) post-cardiac surgery with a good left ventricular ejection fraction without significant co-morbidity. The final decision for PACU-classification is taken by the responsible anaesthesiologist and intensivist in close collaboration with the cardiothoracic surgeon performing the operation, as well as the cardiologist.

SUMMARY:
Determining fluid responsiveness in critically ill patients by measuring mean systemic filling pressure on the intensive care unit.

DETAILED DESCRIPTION:
The assessment of the cardiovascular state in critically ill patients is subject to difficulties in terms of the fact that several hemodynamic parameters, for example mean arterial blood pressure (MAP) and cardiac output (CO) supply insufficient information about the circulating volume and cardiac performance. There is a clinical need to adequate determination of intravascular volume status and therefore reliable predictors of fluid responsiveness are highly relevant. However, in determining the fluid status of a patient, the lack of appreciation of the venous side of the circulation persists today, which is greatly due to the inability to appropriately assess the venous side of the circulation. The importance of the venous part of the circulation is moreover reflected by the fact that an increase in venous resistance does reduce CO many times more than a similar increase in arterial resistance. Mean systemic filling pressure (Pms), which is defined as the pressure equal to the pressure which would be measured if the heart should suddenly stop pumping and all (arterial and venous) the pressures in the entire circulatory system should be brought to equilibrium instantaneously, is a good, complete and reliable reflection of the total intravascular fluid compartment. Passive leg raising (PLR) represents a "self-volume challenge" that predicts preload responsiveness and the transient hemodynamic changes on venous return can be directly monitored in ventilated patients, provided that there is an intact circulation, in order to test the amount of volume responsiveness.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be older than 18 years, and must be equipped with a pulse-contour cardiac output system with a central venous catheter. Patients will be subsequently connected to the hemodynamic monitoring device Navigator™. In those patients with clinical signs of inadequate tissue perfusion, passive leg raising and standardized fluid challenge will be performed.

Exclusion Criteria:

* Patients with assist devices (e.g. intra aortic balloon pump, Impella®, ECMO), patients with arrhythmias (either atrial of ventricular) will be excluded from the study. Also, patients with inguinal impairment or contraindications for a passive leg raising will be excluded (such as deep venous thrombosis or elastic compression stocking), head trauma, an increase intra-abdominal pressure suspected by clinical context and examination as well as patients with absolute contraindications for fluid challenge.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Coronary artery bypass grafting, aortic valve replacement and septic shock patients
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Mean systemic filling pressure (Pms) | 1 hour
  An increase in mean systemic filling pressure after (self)volume-challenge indicating volume responsiveness of the patient

SECONDARY OUTCOMES:
Heart performance (eH) | 1 hour
  Quotient of driving pressure of venous return in mmHg

OTHER OUTCOMES:
Secondary hemodynamic parameters | 1 hour
  Heart Rate
Secondary hemodynamic parameters | 1 hour
  Mean Arterial Blood Pressure
Secondary hemodynamic parameters | 1 hour
  Cardiac Index
Secondary hemodynamic parameters | 1 hour
  Central Venous Pressure
Secondary hemodynamic parameters | 1 hour
  Systemic Vascular Resistance
Secondary hemodynamic parameters | 1 hour
  Pulse Pressure Variation
Secondary hemodynamic parameters | 1 hour
  Pulmonary Vascular Permeability Index
Secondary hemodynamic parameters | 1 hour
  Plethysmographic Oxygen Saturation
Secondary hemodynamic parameters | 1 hour
  Delivery of Oxygen Index
Secondary hemodynamic parameters | 1 hour
  Mechanical Ventilation Settings
Secondary hemodynamic parameters | 1 hour
  End-tidal CO2
Secondary hemodynamic parameters | 1 hour
  Peripheral Temperature

CONTACTS AND LOCATIONS:
Overall Officials: Jan Bakker, PhD, Study Chair — Erasmus University Hospital Rotterdam The Netherlands
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: No
No, data remain anonymized within hospital and property of PI.

REFERENCES:
- [Background] Parkin WG, Leaning MS. Therapeutic control of the circulation. J Clin Monit Comput. 2008 Dec;22(6):391-400. doi: 10.1007/s10877-008-9147-7. Epub 2008 Nov 12. PMID 19002596
- [Background] Lansdorp B, Lemson J, van Putten MJ, de Keijzer A, van der Hoeven JG, Pickkers P. Dynamic indices do not predict volume responsiveness in routine clinical practice. Br J Anaesth. 2012 Mar;108(3):395-401. doi: 10.1093/bja/aer411. Epub 2011 Dec 20. PMID 22185905
- [Background] Michard F, Teboul JL. Predicting fluid responsiveness in ICU patients: a critical analysis of the evidence. Chest. 2002 Jun;121(6):2000-8. doi: 10.1378/chest.121.6.2000. PMID 12065368
- [Background] Monnet X, Rienzo M, Osman D, Anguel N, Richard C, Pinsky MR, Teboul JL. Passive leg raising predicts fluid responsiveness in the critically ill. Crit Care Med. 2006 May;34(5):1402-7. doi: 10.1097/01.CCM.0000215453.11735.06. PMID 16540963
- [Background] Keller G, Desebbe O, Benard M, Bouchet JB, Lehot JJ. Bedside assessment of passive leg raising effects on venous return. J Clin Monit Comput. 2011 Aug;25(4):257-63. doi: 10.1007/s10877-011-9303-3. Epub 2011 Sep 24. PMID 21948105
- [Background] Maas JJ, Geerts BF, van den Berg PC, Pinsky MR, Jansen JR. Assessment of venous return curve and mean systemic filling pressure in postoperative cardiac surgery patients. Crit Care Med. 2009 Mar;37(3):912-8. doi: 10.1097/CCM.0b013e3181961481. PMID 19237896
- [Background] Anderson RM, Fritz JM, O'Hare JE. The mechanical nature of the heart as a pump. Am Heart J. 1967 Jan;73(1):92-105. doi: 10.1016/0002-8703(67)90313-4. No abstract available. PMID 6016029
- [Background] Rothe CF. Mean circulatory filling pressure: its meaning and measurement. J Appl Physiol (1985). 1993 Feb;74(2):499-509. doi: 10.1152/jappl.1993.74.2.499. PMID 8458763
- [Background] GUYTON AC, ABERNATHY B, LANGSTON JB, KAUFMANN BN, FAIRCHILD HM. Relative importance of venous and arterial resistances in controlling venous return and cardiac output. Am J Physiol. 1959 May;196(5):1008-14. doi: 10.1152/ajplegacy.1959.196.5.1008. No abstract available. PMID 13649920
- [Background] GUYTON AC, POLIZO D, ARMSTRONG GG. Mean circulatory filling pressure measured immediately after cessation of heart pumping. Am J Physiol. 1954 Nov;179(2):261-7. doi: 10.1152/ajplegacy.1954.179.2.261. No abstract available. PMID 13218155
- [Background] GUYTON AC, LINDSEY AW, KAUFMANN BN. Effect of mean circulatory filling pressure and other peripheral circulatory factors on cardiac output. Am J Physiol. 1955 Mar;180(3):463-8. doi: 10.1152/ajplegacy.1955.180.3.463. No abstract available. PMID 14376522
- [Background] GUYTON AC, LINDSEY AW, ABERNATHY B, RICHARDSON T. Venous return at various right atrial pressures and the normal venous return curve. Am J Physiol. 1957 Jun;189(3):609-15. doi: 10.1152/ajplegacy.1957.189.3.609. No abstract available. PMID 13458395
- [Background] Parkin WG. Volume state control - a new approach. Crit Care Resusc. 1999 Sep;1(3):311-21. PMID 16603021
- [Background] Pellegrino VA, Mudaliar Y, Gopalakrishnan M, Horton MD, Killick CJ, Parkin WG, Playford HR, Raper RF. Computer based haemodynamic guidance system is effective and safe in management of postoperative cardiac surgery patients. Anaesth Intensive Care. 2011 Mar;39(2):191-201. doi: 10.1177/0310057X1103900207. PMID 21485666
- [Background] Jansen JR, Maas JJ, Pinsky MR. Bedside assessment of mean systemic filling pressure. Curr Opin Crit Care. 2010 Jun;16(3):231-6. doi: 10.1097/MCC.0b013e3283378185. PMID 20168223
- [Background] Maas JJ, Pinsky MR, Geerts BF, de Wilde RB, Jansen JR. Estimation of mean systemic filling pressure in postoperative cardiac surgery patients with three methods. Intensive Care Med. 2012 Sep;38(9):1452-60. doi: 10.1007/s00134-012-2586-0. Epub 2012 May 15. PMID 22584797
- [Background] Lang RM, Bierig M, Devereux RB, Flachskampf FA, Foster E, Pellikka PA, Picard MH, Roman MJ, Seward J, Shanewise JS, Solomon SD, Spencer KT, Sutton MS, Stewart WJ; Chamber Quantification Writing Group; American Society of Echocardiography's Guidelines and Standards Committee; European Association of Echocardiography. Recommendations for chamber quantification: a report from the American Society of Echocardiography's Guidelines and Standards Committee and the Chamber Quantification Writing Group, developed in conjunction with the European Association of Echocardiography, a branch of the European Society of Cardiology. J Am Soc Echocardiogr. 2005 Dec;18(12):1440-63. doi: 10.1016/j.echo.2005.10.005. No abstract available. PMID 16376782
- [Background] Oren-Grinberg A. The PiCCO Monitor. Int Anesthesiol Clin. 2010 Winter;48(1):57-85. doi: 10.1097/AIA.0b013e3181c3dc11. No abstract available. PMID 20065727
- [Background] Bakker J, Damen J, van Zanten AR, Hubben JH; Protocollencommissie Nederlandse Vereiniging voor Intensive Care. [Admission and discharge criteria for intensive care departments]. Ned Tijdschr Geneeskd. 2003 Jan 18;147(3):110-5. Dutch. PMID 12577770
- [Background] Jabot J, Teboul JL, Richard C, Monnet X. Passive leg raising for predicting fluid responsiveness: importance of the postural change. Intensive Care Med. 2009 Jan;35(1):85-90. doi: 10.1007/s00134-008-1293-3. Epub 2008 Sep 16. PMID 18795254
- [Background] Jolly SS, Yusuf S, Cairns J, Niemela K, Xavier D, Widimsky P, Budaj A, Niemela M, Valentin V, Lewis BS, Avezum A, Steg PG, Rao SV, Gao P, Afzal R, Joyner CD, Chrolavicius S, Mehta SR; RIVAL trial group. Radial versus femoral access for coronary angiography and intervention in patients with acute coronary syndromes (RIVAL): a randomised, parallel group, multicentre trial. Lancet. 2011 Apr 23;377(9775):1409-20. doi: 10.1016/S0140-6736(11)60404-2. Epub 2011 Apr 4. PMID 21470671